CLINICAL TRIAL: NCT05693220
Title: The Sperm Preparation Prior to Intrauterine Insemination Study (PIoUS)
Brief Title: Sperm Preparation Prior to Intrauterine Insemination Study
Acronym: PIoUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-36913
Record Dates: First submitted 2022-12-09; First posted 2023-01-20 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Infertility; Infertility Secondary; Infertility Unexplained; Anovulation; Fertility Disorders; Reproductive Issues
Keywords: Intrauterine Insemination; Insemination; Fertility; Infertility
MeSH Terms: conditions — Infertility; Anovulation | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Density gradient centrifugation (Active Comparator): Patients will undergo sperm preparation by density gradient centrifugation
  Interventions: Other: Density gradient centrifugation
- Zymot sperm separation device (Active Comparator): Patients will undergo sperm preparation by the Zymot sperm separation device
  Interventions: Device: Zymot Multi sperm separation device

INTERVENTIONS:
Device: Zymot Multi sperm separation device — Sperm preparation with Zymot Multi sperm preparation device
  Arms: Zymot sperm separation device
Other: Density gradient centrifugation — Sperm preparation with density gradient centrifugation
  Arms: Density gradient centrifugation

SUMMARY:
This is a randomized controlled trial comparing density gradient centrifugation and microfluidic sperm sorting in patients undergoing intrauterine insemination to evaluate cumulative pregnancy outcomes.

DETAILED DESCRIPTION:
Study participants will be randomized to either standard sperm preparation (density gradient centrifugation) versus sperm preparation with the Zymot Multi sperm preparation device for their three month intrauterine insemination treatment course. Patients will follow standard treatment plans designed by their fertility physician and will be followed until referred for prenatal care at 8-10 weeks of pregnancy to determine pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing intrauterine insemination
* Patient assigned female at birth with age <41

Exclusion Criteria:

* Any significant disease or psychiatric disorder that would interfere with the consenting process
* Prior intrauterine insemination
* Use of frozen donor sperm
* Non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative clinical pregnancy rate | 3 treatment cycles, an average of 5 months
  The clinical pregnancy rate by treatment group over the course of IUI treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gode F, Bodur T, Gunturkun F, Gurbuz AS, Tamer B, Pala I, Isik AZ. Comparison of microfluid sperm sorting chip and density gradient methods for use in intrauterine insemination cycles. Fertil Steril. 2019 Nov;112(5):842-848.e1. doi: 10.1016/j.fertnstert.2019.06.037. Epub 2019 Sep 19. PMID 31543253
- [Background] Quinn MM, Jalalian L, Ribeiro S, Ona K, Demirci U, Cedars MI, Rosen MP. Microfluidic sorting selects sperm for clinical use with reduced DNA damage compared to density gradient centrifugation with swim-up in split semen samples. Hum Reprod. 2018 Aug 1;33(8):1388-1393. doi: 10.1093/humrep/dey239. PMID 30007319